CLINICAL TRIAL: NCT06006741
Title: Universal CAR-T Cells for the Treatment of Multiple Myeloma
Brief Title: Universal CAR-T Cells Targeting Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-23003
Record Dates: First submitted 2023-08-08; First posted 2023-08-23 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Multiple Myeloma in Remission
Keywords: Universal CART; multiple myelomachimeric antigen BCMA CD38 CD56 CD138 CD19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Universal CART cells to treat MM (Experimental)
  Interventions: Biological: MM-specific universal CAR T cells

INTERVENTIONS:
Biological: MM-specific universal CAR T cells — Infusion of MM-specific universal CAR T cells

SUMMARY:
The aim of this study is to assess the feasibility, safety and efficacy of universal CAR T cells targeting multiple myeloma. Another goal of the study is to learn more about the persistence and function of the universal CAR T cells in the body.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a malignancy of the plasma cells, which remains a clinical challenge despite advanced therapeutic interventions including novel molecular therapies and stem cell transplantation (SCT).

CAR-T therapy has proven to be a revolutionary treatment for hematological malignancies, but its manufacture is still limited by the high cost, and a long preparation time that is not conducive to timely treatment of patients. In addition, many MM patients suffer from long-term bone marrow suppression caused by tumor growth or prolonged and intense chemotherapies, resulting in exhaustion, aging and functional defects of autologous T cells, which substantially affect the quality of CAR-T cells and the clinical efficacy. The universal CAR-T cells could overcome many of the above problems.

By using universal type of CAR-T cells, the product can be supplied off-the-shelf without being customized from individual patients. In addition, the immediate availability means that patients under severe bone marrow suppression may get a chance to be treated with CAR-T cells to achieve disease remission. In addition, those patients who suffer from long-term immunosuppression due to tumor microenvironment or myelosuppressive chemotherapy would have the option of treatment with the universal CAR-T cells.

The purpose of this study is to assess the feasibility, safety and efficacy of several 4SCAR designs including BCMA, CD138, CD38 and CD19-specific universal CAR-T products targeting MM. Another goal is to learn more about the function of these universal CAR T cells and their persistency in the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed multiple myeloma failed curative treatment options (including autologous or allogeneic SCT).
2. Complete remission (CR) cannot be achieved after at least 2 prior therapy regimens.
3. High risk MM in CR1 or CR2 and not eligible for SCT because of age or comorbid diseases.
4. Less than 1 year between last chemotherapy and progression (i.e. most recent progression free interval < 1 year).
5. Relapsed after prior autologous or allogenic SCT with residual disease after at least 1 prior therapy and not eligible for allogeneic SCT.
6. Residual disease after primary therapy and not eligible for ASCT
7. Expected survival > 12 weeks• Creatinine < 2.5 mg/dl• ALT (alanine aminotransferase)/AST (aspartate aminotransferase) < 3x normal
8. Bilirubin < 2.0 mg/dl
9. Any relapse after prior SCT is eligible regardless of other prior therapy
10. Adequate venous access for apheresis, and no other contraindications for leukapheresis
11. Voluntary informed consent is signed

Exclusion Criteria:

1. Pregnant or lactating women
2. Uncontrolled active infection
3. Active hepatitis B or hepatitis C infection
4. Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary.
5. Previous related CAR-T cell therapy
6. Any uncontrolled active medical disorder that would preclude participation
7. HIV infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-31 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with treatment related adverse effect | 6 months
  percentage of participants with treatment-related adverse events, as assessed by physical examination, vital signs, standard clinical lab tests.

SECONDARY OUTCOMES:
Anti-tumor activity of the universal 4SCAR-T cells after infusion | 3 months
  CART cells in the peripheral blood of patients will be measured by qPCR on Day 7, 14, 21, 28, 60 and 90 after infusion.
Anti-tumor activity of fourth generation universal CAR-T cells in patients with relapsed or refractory MM | 1 year
  Objective response, such as complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD) will be assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Geno-Immune Medical Institute, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No